CLINICAL TRIAL: NCT07147296
Title: ARC-IM System to Manage Symptomatic Blood Pressure Instability Secondary to Chronic Spinal Cord Injury
Acronym: Empower BP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ONWARD Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ONWD-IM-001
Record Dates: First submitted 2025-08-14; First posted 2025-08-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries; Blood Pressure Disorders
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: Randomized and sham-controlled study consisting of a 3-month double-blinded phase followed by a 21-month open-label phase
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active Group (Experimental): ARC-IM System with active stimulation since day 0
  Interventions: Procedure: ARC-IM System Implantation; Device: ARC-IM Therapy (active)
- Sham Group (Sham Comparator): ARC-IM System without active stimulation before the open-label phase of the study (3 month post-implant)
  Interventions: Procedure: ARC-IM System Implantation; Device: ARC-IM Therapy (sham)

INTERVENTIONS:
Procedure: ARC-IM System Implantation — Implantation of the ARC-IM Thoracic Lead in the epidural space and ARC-IM Neurostimulator
Device: ARC-IM Therapy (active) — The ARC-IM System is programmed since day 0 to deliver active electrical spinal cord stimulation at the low thoracic level for the management of symptomatic blood pressure instability in people with chronic spinal cord injury
  Arms: Active Group
Device: ARC-IM Therapy (sham) — The ARC-IM System is programmed at month 3 to deliver active electrical spinal cord stimulation (after 3 months of sham stimulation) at the low thoracic level for the management of symptomatic blood pressure instability in people with chronic spinal cord injury
  Arms: Sham Group

SUMMARY:
Empower BP is a pivotal, interventional, multicenter, prospective, randomized, sham-controlled double-blinded study to evaluate the safety and effectiveness of the ARC-IM System in managing symptomatic blood pressure instability in individuals with chronic SCI (>1 year after SCI).

The primary effectiveness outcome will be evaluated through subject-reported ADFSCI and seated blood pressure assessments at 3 months post-implant.

Following a baseline screening period and the surgical implantation of the ARC-IM System, subjects will be randomized with a 2:1 ratio into an active or control arm for 3 months. All the subjects will undergo therapy activation sessions (active or sham) within 21 days of the surgical implant and will then commence independent at-home use of ARC-IM Therapy. At the 3 Month timepoint, after all assessments are conducted, all subjects will transition to the open-label period in order to receive the active version of the ARC-IM System in an open-label fashion. All subjects will undergo therapy programming sessions following Month 3.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or above, and no older than 75 years at the time of enrollment.
2. Clinical evidence of Orthostatic Hypotension (blood pressure drop of 20mmHg systolic or 10mmHg diastolic) measured during Head Up Tilt Table assessment (HUTT, within 10 minutes) with current standard of care if any. 2 out of 3 tests must meet OH criteria.
3. Clinical evidence of sustained hypotension (average systolic Blood pressure ≤ 110 mmHg) when measured each minute for 10 minutes while seated and in the absence of supportive compressive garments and medication.
4. Evidence of symptomatic hypotension as determined by a non-zero OHSA total score
5. A Spinal cord injury at the neurologic level between C2 and T6 inclusive.
6. American Spinal Injury Association (ASIA) Impairment Scale (AIS) classification A, B, C, or D.
7. Traumatic (non-progressive) chronic spinal cord injury with minimum 12 months post-injury prior to study entry.
8. Average A-P diameter of the sponal canal ≥ 13 mm, measured on MRI at the disc space at level(s) planned for implantation
9. Stable medical, physical, and psychological condition as considered by the investigators.
10. Stable dose of blood pressure medication for 30-days prior to enrollment into the study . Stability will be defined as no changes to medication regimens based on treating physician instructions.
11. Subjects who are on long-term antihypertensive treatment must discontinue these medications no less than 30 days prior to enrollment in the study. This requirement does not apply to antihypertensive agents administered for the acute management of autonomic dysreflexia (AD)
12. If the subject requires daily continuous support from a personal caregiver, the presence of a caregiver during the study visits is mandatory.
13. Willing and able to provide informed consent.
14. Stated willingness to comply with all study procedures and availability for the duration of the study.
15. Willing and able to comply with the instructions for use, operate the study devices, and comply with this clinical investigation plan

Exclusion Criteria:

1. Subject has an autoimmune etiology of spinal cord dysfunction/injury.
2. Subject has diseases and conditions that would increase the morbidity and mortality of the surgical procedures required by the study.
3. Subject has a history of physiologic hypotension prior to SCI
4. Subject has a history of unexpected blood pressure instability related to medications
5. Inability to withhold antiplatelet/anticoagulation agents perioperatively.
6. History of myocardial infarction or cerebrovascular event within the past 6 months. or
7. History of chronic/recurrent severe cardiac arrythmias (e.g., ventricular tachycardia, ventricular fibrillation, third degree atrioventricular block)
8. Evidence of clinically significant underlying cardiac conditions on Holter monitoring performed at screening including but not limited to arrhythmias (e.g., atrial fibrillation, ventricular tachycardia),
9. Evidence of ischemic changes or prolonged QT interval (QTc > of 450 ms for males and 470 ms for females) identified on EKG during screening,
10. Subjects with a known diagnosis of heart failure, including but not limited to New York Heart Association (NYHA) Class I-IV, or with evidence of clinically significant left ventricular dysfunction (ejection fraction < 40%) as determined by echocardiogram during screening or within the past 6 months,
11. Current renal/kidney, hepatic, or other concomitant disorders deemed severe by the Investigator including those ones that could be linked to severe autonomic dysreflexia.
12. Requires continuous ventilator support.
13. Imaging (MRI, CT, X-ray) findings within the last 12 months that contraindicate lead placement
14. Known allergic reaction to implanted materials
15. Requires continuous/frequent/any transcutaneous spinal cord stimulation treatment.
16. Has any active implanted medical device (e.g. baclofen pump, pacemaker).
17. Inability to receive a pre-operative MRI.
18. Female subject who is pregnant, breastfeeding or planning to become pregnant or breastfeed. Women of child-bearing potential must have a negative pregnancy test completed at baseline visit per site standard test.
19. Presence of pressure sore at time of screening or baseline graded stage 3 or 4 .
20. Subject is enrolled or intends to participate in another clinical drug and/or device study or registry that may interfere with the results of this study, as determined by ONWARD Medical personnel.
21. Presence of other anatomic or comorbid conditions, or other medical, social, or psychologic conditions such as severe uncontrolled neuropathic pain, depression, history of alcohol or substance abuse, history of schizophrenia or psychotic illness, severe personality disorder or other significant psychiatric or cognitive disorders that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements of the clinical investigation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-17 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving a change in the hypotension domain of the ADFSCI short-form questionnaire | 3-months post-implant
  Proportion of subjects achieving a reduction of ≥ 4 points in the hypotension domain of the ADFSCI short-form questionnaire compared to baseline
Proportion of subjects achieving elevation in SBP during seated BP test | 3-months post-implant
  Proportion of subjects achieving an elevation of ≥ 10 mmHg in systolic blood pressure during the seated BP test with stimulation ON compared to stimulation OFF
Incidence of serious adverse device effects | 6-months post-implant
  Description of all Serious Adverse Device Effects from ARC-IM System implant until Month 6

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Craig Hospital, Englewood, Colorado
  - UofL Health - Frazier Rehabilitation Institute, Louisville, Kentucky
  - Spaulding Rehabilitation, Cambridge, Massachusetts
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No